CLINICAL TRIAL: NCT05358353
Title: A Prospective Single-Arm Multicenter StuDy of the BarE TEmporary SPur StEnt System foR the tREatment of Vascular Lesions Located in the infrapoplitEal Arteries beLow the Knee (DEEPER REVEAL)
Acronym: DEEPER REVEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ReFlow Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-007
Record Dates: First submitted 2022-04-15; First posted 2022-05-03 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Arterial Disease; Critical Limb Ischemia
Keywords: Peripheral Arterial Disease; Critical Limb Ischemia; Infrapopliteal Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Bare Temporary Spur Stent System (Experimental): Treatment with the Temporary Bare Spur Stent System (Spur Stent System).
  Interventions: Device: Bare Temporary Spur Stent System

INTERVENTIONS:
Device: Bare Temporary Spur Stent System — Treatment of qualifying infrapopliteal arteries with the Bare Temporary Spur Stent System, in subjects with critical limb ischemia.

SUMMARY:
This is a prospective, multicenter, single arm study designed to evaluate the safety and efficacy of the Temporary Bare Spur Stent System (Spur Stent System).

ELIGIBILITY:
Pre-Procedure Inclusion Criteria:

1. Subject willing and able to provide informed consent and able to comply with the study protocol and follow up. Subjects who are unable to sign due to a physical limitation may have a witness, including a family member, sign on their behalf.
2. Life expectancy greater than 1 year in the investigator's opinion.
3. Male or non-pregnant female ≥18 years of age at time of consent.
4. Subjects must have chronic (greater than 14 days) symptoms of limb ischemia, determined by clinical symptoms of Rutherford class 4-5, rest pain (R 4), and/or minor tissue loss (R5), that in the opinion of the investigator are not amenable to conservative medical therapy and require endovascular intervention for alleviation of symptoms and tissue preservation.
5. For subjects with bilateral disease, planned treatment of the contralateral limb must either be performed greater than or equal to 3 days prior to the index procedure or greater than or equal to 7 days following the index procedure.

Angiographic Inclusion Criteria:

1. Stenotic, restenotic, or occlusive lesions located in the infrapopliteal vessels, with target lesion that can be successfully crossed via the true lumen with a guidewire (no subintimal crossing).
2. Iliac, SFA and popliteal inflow lesions can be treated using standard of care during the index procedure or greater than or equal to 3 days prior.

   Note:
   1. Inflow lesions treated intraprocedure must be treated first, prior to consideration of treatment of infrapopliteal lesions.
   2. Treatment of in-stent restenosis in inflow treatment is permitted, provided that stents are not fractured or otherwise compromised.
   3. Distal embolic protection is strongly encouraged in cases where atherectomy is used.
   4. Inflow lesions must have a healthy vessel segment of greater than 30 mm between the study lesion and the treated segment, defined as less than 50% stenosis without aneurysmal segments.
   5. Inflow treatment must be successful, prior to treatment of the target lesion, resulting in stenosis less than or equal to 30%, without resulting flow limiting dissection, thrombus, or aneurysm by angiography.
3. Target vessel(s) reconstitute(s) at or above the ankle, with the target treated segment ending at least 10 mm above the ankle joint.

   Note:
   1. If the anterior tibial or posterior tibial arteries are treated, there must be inline flow to the foot.
   2. If the peroneal artery is treated, there must be at least one collateral supplying the foot.
   3. In all cases, patent runoff (no lesions with greater than 50% stenosis) must be present via the dorsalis pedis and/or plantar arteries
4. Target lesion must be located in the tibial arteries. If vessel sizing remains appropriate, treatment may extend into the distal popliteal (P3) segment.
5. Target vessel reference diameter is measured to be between 2.5 to 4.5 mm in diameter assessed by one of the following methods after successful completion of guidewire crossing of the lesion site:

   1. Intravascular Ultrasound (IVUS) (primary)
   2. Visual estimate using Angiography (secondary)
6. Target lesion length is less than or equal to 210mm in length. Tandem lesions that are less than or equal to 4 cm should be treated as one lesion. Multiple discrete lesions may be treated provided cumulative length is less than or equal to 210 mm.
7. Successful pre-dilatation of the target lesion defined as resulting in stenosis less than or equal to 50% and/or inner lumen diameter greater than or equal to 2.0 mm in diameter, without resulting flow limiting dissection, thrombus, or aneurysm by angiography prior to the insertion of the Bare Temporary Spur Stent System.
8. Only one limb and one contiguous vessel may be enrolled per subject. If required, a second modality may be used for treatment in the non-target infrapopliteal vessel.

   Note:
   1. Distal embolic protection is strongly recommended in cases using atherectomy.
   2. Treatment of the target vessel/lesion may be performed only if treatment of the non-target lesion is successful without resulting flow limiting (Type D or greater) dissection, thrombus, or aneurysm by angiography.
   3. Treatment of non-target lesions must be parallel to, and not contiguous with, the target lesion.
9. If pre-screening with duplex ultrasound, angiography, CTA, or MRA has been performed less than or equal to 365 days prior to the procedure, intra-procedure angiography of the aorto-iliac vasculature is not required, however, the femoropopliteal inflow must still be imaged using angiography during the index procedure.
10. Retrograde access (in the infrapopliteal arteries) is permitted for lesion crossing; however, the Bare Temporary Spur Stent System must be deployed from antegrade (above the knee, either ipsilateral or contralateral) access.

Pre-procedure Exclusion Criteria:

1. Subject unwilling or unlikely to comply with the 1-year duration of the study in the opinion of the investigator.
2. Subject is pregnant or planning to become pregnant during the course of the trial.
3. Subject has an active systemic infection that is not controlled at the time of the procedure, including septicemia or bacteremia.
4. Subject has osteomyelitis proximal to the phalanges. Osteomyelitis in the digit(s) of the target foot is permitted.
5. Wounds must be confined to the foot below the ankle. Heel wounds are excluded.
6. Planned major (above the ankle) amputation of the target limb. A planned or previous minor (trans metatarsal amputation or digit amputation) is permitted.
7. Recent myocardial infarction or stroke less than 90 days prior to the index procedure.
8. Symptomatic acute heart failure NYHA class III or greater.
9. Impaired renal function (eGFR less than or equal to 25 mL/min) within 30 days of procedure or end stage renal disease on dialysis.
10. Inability to tolerate dual antiplatelet and/or anticoagulation therapy.
11. Known allergies or sensitivities to heparin, antiplatelet drugs, other anticoagulant therapies which could not be substituted, or an allergy to contrast media that cannot be adequately pre-treated prior to the index procedure.
12. The subject is currently enrolled in another investigational device or drug trial that interferes with the study endpoints.
13. Known allergy to nitinol or nickel.
14. Bypass surgery of the target vessel(s). Prior bypass above the level of the infrapopliteal arteries is permitted.

Angiographic Exclusion Criteria

1. Target lesion is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion. Inflow must also be free of aneurysmal segments.
2. Fractured or otherwise compromised stents in the target vessel or inflow vessel.
3. In-stent restenosis in the target vessel.
4. Previous treatment of inflow lesions performed less than or equal to 7 days prior to the index procedure.
5. Previous treatment of the target vessel less than or equal to 90 days prior to index procedure.
6. Angiographic evidence of thrombus within target limb.
7. Extremely severe calcification that, in the investigator's opinion, would not be amenable to PTA.
8. Type D dissections or greater incurred during CTO crossing (see Appendix I for definitions).
9. Significant (greater than or equal to 50%) stenosis of inflow arteries or unsuccessful treatment of inflow lesions.
10. Distance from access to lesion is too long for a 135 cm working length of the Bare Temporary Spur Stent System catheter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2025-05-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (48):
  - St. Bernards Heart and Vascular, Jonesboro, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - University of California, Irvine Health, Orange, California
  - Vascular & Interventional Specialist of Orange County, Orange, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - Vascular Care Connecticut (site) / Vascular Breakthroughs (research support), Darien, Connecticut
  - Southern CT Vascular Center, Shelton, Connecticut
  - Palm Beach Heart and Vascular, Boynton Beach, Florida
  - Bradenton Cardiology, Bradenton, Florida
  - Delray Medical Center, Delray Beach, Florida
  - First Coast Cardiovascular Institute, Fleming Island, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Surgical Specialists of Ocala, Ocala, Florida
  - Ansaarie Cardiac & Endovascular Center of Excellence, Palatka, Florida
  - Coastal Vascular and Interventional Center, Pensacola, Florida
  - Guardian Research, Winter Park, Florida
  - Rush University, Chicago, Illinois
  - Midwest Cardiovascular Institute, Naperville, Illinois
  - Community Healthcare Systems, Munster, Indiana
  - UnityPoint Health Trinity Bettendorf Hospital, Bettendorf, Iowa
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Cardiovascular Institute of the South, Lafayette, Louisiana
  - Ochsner Health, New Orleans, Louisiana
  - Massachusetts General Hospital, Somerville, Massachusetts
  - Vascular Care Group (site) / Vascular Breakthroughs (research support), Wellesley, Massachusetts
  - Advanced Cardiac and Vascular Centers for Amputation Prevention, Grand Rapids, Michigan
  - Advanced Vascular Surgery, Kalamazoo, Michigan
  - Eastlake Cardiovascular PC, Roseville, Michigan
  - University of Missouri, Columbia, Missouri
  - Mercy South, St Louis, Missouri
  - Advanced Heart and Vascular Institute of Hunterdon, Flemington, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Novant Health Heart & Vascular Institute, Matthews, North Carolina
  - Sunrise Vascular, Murphy, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Health, Columbus, Ohio
  - Lankenau Institute for Medical Research, Bryn Mawr, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Prisma Health, Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac and Vascular Institute, Corpus Christi, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - El Paso Cardiology Associates, El Paso, Texas
  - Texas Tech University Health Sciences Center, Odessa, Texas
  - Sentara Norfolk General, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bare Temporary Spur Stent System
Started | 130
Completed | 105
Not Completed | 25

BASELINE CHARACTERISTICS:
Arm/Group | Bare Temporary Spur Stent System
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 102
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 130

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint: Percentage of Participants With Technical Success of the Bare Temporary Spur Stent
Description: Technical Success is defined as <30% residual stenosis in subjects treated with the Bare Temporary Spur Stent System
Time Frame: At the end of the Index Procedure
Measure: Number; unit: percentage of participants
Arm/Group | Bare Temporary Spur Stent System
Number analyzed (Participants) | 130
percentage of participants | 99.2

2. Primary Outcome: Co-Primary Safety Endpoint: Percentage of Patients With no Major Adverse Limb Event (MALE) or Peri-operative Death (POD) at 30 Days Post Procedure
Description: Number of participants with freedom from the occurrence of major adverse limb events (MALE) [evaluated at 30 days post procedure] and peri-operative death (POD) [defined as all-cause mortality within 30 days post procedure].
  MALE is defined as:
  * Above-the-ankle amputation of the index limb
  * Major reintervention (new bypass graft, jump/interposition graft revision, or thrombectomy/thrombolysis) of the index limb involving the infrapopliteal arteries.
Time Frame: 30 days post procedure
Measure: Number; unit: percentage of participants
Arm/Group | Bare Temporary Spur Stent System
Number analyzed (Participants) | 130
percentage of participants | 96.7

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Bare Temporary Spur Stent System
All-Cause Mortality (participants affected / at risk) | 3/130
Serious Adverse Events (participants affected / at risk) | 30/130
Other Adverse Events (participants affected / at risk) | 53/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bare Temporary Spur Stent System (N=130)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Acute MI (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (2)
Peripheral swelling (Cardiac disorders) | 1 (1)
Ventricular tachycardic (Cardiac disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Gangrene (Infections and infestations) | 2 (2)
Osteomyelitis (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gangrene (Skin and subcutaneous tissue disorders) | 1 (1)
Foot amputation (Surgical and medical procedures) | 2 (2)
Toe amputation (Surgical and medical procedures) | 3 (3)
Peripheral revascularization (Surgical and medical procedures) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 4 (4)
Arterial occlusive disease (Vascular disorders) | 2 (2)
Artery dissection (Vascular disorders) | 1 (1)
Carotid artery stenosis (Vascular disorders) | 1 (1)
Epistaxis (Vascular disorders) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (2)
Hypertensive crisis (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral ischemia (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bare Temporary Spur Stent System (N=130)
Acute Kidney Injury (Metabolism and nutrition disorders) | 1 (1)
Artery Dissection (Vascular disorders) | 3 (3)
Amputation (Surgical and medical procedures) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Food Poisoning (Infections and infestations) | 1 (1)
Foot Amputation (Surgical and medical procedures) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Limb Injury (Injury, poisoning and procedural complications) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathic Arthropathy (Nervous system disorders) | 1 (1)
Oedema Peripheral (Cardiac disorders) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1)
Oedema Peripheral (Metabolism and nutrition disorders) | 1 (1)
Osteomyelitis (Infections and infestations) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1)
Peripheral Artery Dissection (Vascular disorders) | 2 (3)
Peripheral Swelling (General disorders) | 1 (1)
Peripheral Venous Disease (Vascular disorders) | 1 (1)
Procedural Pain (General disorders) | 1 (1)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Sars-CoV-2 test positive (Investigations) | 1 (1)
Serratia Infection (Infections and infestations) | 1 (1)
Skin Wound (Injury, poisoning and procedural complications) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1)
Subcutaneous Abscess (Skin and subcutaneous tissue disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Toe Amputation (Surgical and medical procedures) | 2 (2)
Vasospasm (Vascular disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wound (Skin and subcutaneous tissue disorders) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT05358353/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT05358353/ICF_001.pdf